CLINICAL TRIAL: NCT02079896
Title: Safety, PK/PD, and Efficacy of NOX-H94 in Dialysis Patients With ESA-hyporesponsive Anemia: A Randomized, Double Blind, Placebo Controlled Parallel Group Study With a Single Blind Cross-over Group
Brief Title: Lexaptepid Pegol (NOX-H94) in ESA-hyporesponsive Anemia in Dialysis Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNOXH94C301; 2013-003585-14 (EudraCT Number)
Record Dates: First submitted 2014-02-28; First posted 2014-03-06 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Anemia; End Stage Renal Disease
Keywords: Dialysis
MeSH Terms: conditions — Anemia; Kidney Failure, Chronic | interventions — NOX-H94

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Single dose cross-over pilot (Experimental): Single dose of lexaptepid pegol (NOX-H94) cross-over with single dose of placebo
  Interventions: Drug: Lexaptepid pegol (NOX-H94); Drug: Placebo
- Control (Placebo Comparator): Twice weekly doses of placebo, 9 total
  Interventions: Drug: Placebo
- Lexaptepid pegol (NOX-H94) (Experimental): Twice weekly doses of lexaptepid pegol (NOX-H94), 9 total
  Interventions: Drug: Lexaptepid pegol (NOX-H94)

INTERVENTIONS:
Drug: Lexaptepid pegol (NOX-H94) — anti-hepcidin L-RNA-aptamer (Spiegelmer)
  Other Names: NOX-H94
  Arms: Lexaptepid pegol (NOX-H94); Single dose cross-over pilot
Drug: Placebo
  Arms: Control; Single dose cross-over pilot

SUMMARY:
Dialysis patients regularly suffer from anemia which may be caused by various contributing factors, alone or in combination, including blood loss, low erythropoietin and iron sequestration. In most patients, the anemia is responsive to treatment with erythropoietin or other erythropoiesis stimulating agents (ESA) alone or in combination with intravenous (i.v.) iron. In about 10% of patients however, the anaemia does not respond appropriately to this standard treatment and high to very high doses of ESA and i.v. iron are used to maintain acceptable hemoglobin concentrations. In these patients, hepcidin was identified as a causative factor leading to anemia of chronic disease with functional iron deficiency and ESA-hyporesponsiveness.

The Spiegelmer lexaptepid pegol (NOX-H94) offers a hepcidin-specific approach to the treatment of anemia of chronic disease. The safety and the activity of lexaptepid pegol are supported by data from healthy subjects and patients with multiple myeloma or lymphoma. The present study in dialysis patients with functional iron deficiency and ESA-hyporesponsiveness is conducted to demonstrate the safety of lexaptepid pegol in this population, to investigate its pharmacokinetic (PK) and pharmacodynamic (PD) profiles and its efficacy in increasing haemoglobin (Hb) in dialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease treated with maintenance hemodialysis.
* Anemia : Hb 7 to 11 g/dL.
* Functional iron deficiency: Transferrin saturation <30%, Ferritin ≥300 ng/mL.
* ESA-hyporesponsiveness with erythropoietin dose ≥12,000 IU/ week.

Exclusion Criteria:

* Treatment with darbepoetin or methoxy-polyethyleneglycol-epoetin.
* Uncontrolled / unstable cardiovascular , peripheral arterial or cerebrovascular disease.
* Congestive heart failure: New York Heart Association Class III or IV.
* Unstable angina, myocardial infarction, percutaneous transluminal coronary angioplasty/stents, or coronary artery bypass grafting <3 months prior screening.
* Any other medical conditions requiring a change in treatment within 4 weeks prior to screening or making study participation unadvisable.
* History of clinically relevant hemolysis and/or blood loss.
* AST, ALT, or bilirubin ≥2.0 times the upper limit of normal.
* Known bone marrow fibrosis.
* Treatment with i.v. iron <4 weeks prior to screening or during the screening period or change in erythropoietin dose during last month.
* Any acute or chronic infection, viral or bacterial within 4 weeks prior to screening or during the screening period considered as systemic infection.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | up to 8 weeks

SECONDARY OUTCOMES:
Pharmacokinetics | Weeks 1, 2, 3, 4, 5, 6, 8
  Peak concentrations, systemic exposure, elimination
Pharmacodynamics | 0 to 48 hours
  Change in serum iron concentrations
Efficacy | Weeks 1, 2, 3, 4, 5, 6, 8
  Change in hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Kai Riecke, MD, Study Director — TME Pharma AG
Locations (10):
- Germany (4):
  - Dialysis Unit, Düsseldorf
  - University Hospital, Halle
  - Hospital, Leipzig
  - Dialysis Unit, Villingen-Schwenningen
- Hospital, Siena, Italy
- United Kingdom (5):
  - Hospital, Swansea, Wales
  - Hospital, Leicester
  - Hospital, London
  - King's College London, London
  - Lister Hospital, Stevenage

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581